CLINICAL TRIAL: NCT01728987
Title: The Significance of Vitamin D Storage in Adipose Tissue
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: study stopped due to Financial problems
Sponsor: University of Tromso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: TromsøEndo-2012-1
Record Dates: First submitted 2012-09-03; First posted 2012-11-20 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cholecalciferol (Active Comparator): vitamin d (cholecalciferol) will be given as a capsule of 20.000 Iu twice a week
  Interventions: Drug: cholecalciferol
- placebo (Placebo Comparator): the placebo capsules are looking identical to the vitamin d capsules and contain medium chain triglycerides and arachis oil
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: cholecalciferol — as in arm description
  Other Names: Dekristol
  Arms: cholecalciferol
Drug: placebo — capsule looking identical to the cholecalciferol capsule
  Arms: placebo

SUMMARY:
The study will examine the role of adipose tissue in vitamin D physiology, particularly its role as a depot. the study is randomized double blind and placebo controlled.

DETAILED DESCRIPTION:
vitamin d versus placebo will be given for 12 months. Biopsies will be taken at baseline and every 6 month for 2 years. Blood samples will be collected every 6th month. the study will thus give information on storage during vitamin d supplementation as well as use of vitamin d fat stores after stopping vitamin D supplementation

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* hypercalcemia
* pregnancy
* women without safe contraception

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
vitamin D in adipose tissue biopsies | 12 months

SECONDARY OUTCOMES:
rate of decline of 25ohd in serum | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: rolf jorde, professor, Principal Investigator — University of Tromsø, Norway
Locations (1):
- University of Tromsø, Tromsø, Tromsø, Norway